CLINICAL TRIAL: NCT04946162
Title: The Use of Tadalafil in Confirmed COVID-19 Pneumonia.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The investigators never completed the IRB application due to decrease in need to conduct the study.
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-63mrx
Record Dates: First submitted 2021-06-28; First posted 2021-06-30 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: COVID; Sars-CoV2; ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: Participants will serve as a self-control, with values recorded pre-medication, 30 minutes after medication administration, and 4 hours after administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tadalafil Group (Experimental): Each patient will be given tadalafil 40 mg one time
  Interventions: Drug: Tadalafil Pill

INTERVENTIONS:
Drug: Tadalafil Pill — Each patient will be given tadalafil 40 mg one time

SUMMARY:
Our goal is to assess the effects of Tadalafil in the setting of confirmed COVID-19 pneumonia. In particular we plan to assess its effects on oxygen saturation, P:F ratio, and mixed central venous oxygen

We plan to recruit all hospitalized patients at Santa Barbara Cottage Hospital with a confirmed COVID19 pneumonia (positive PCR + clinical signs/symptoms of lower respiratory disease) who meet the Berlin definition of ARDS and have access to measure a mixed venous oxygen saturation. For the purposes of obtaining mixed central venous oxygen, all participating patients will already have an internal jugular central venous catheter in place for inclusion in this study. Since all patients will be intubated, their Legally Authorized Representative (LAR) will be approached to discuss the study and asked to participate in the study by an ICU physician, either the attending physician or a medical resident.

Informed consent will be obtained from the LAR by an ICU attending physician or resident involved in the study prior to participation. Patients who meet the above eligibility criteria will have baseline levels of mixed central venous oxygen, oxygen saturation, P:F ratio, blood pressure and PaO2 recorded.

Each patient will then receive Tadalafil 40mg once. The above listed parameters will be monitored again 30 minutes after drug administration and 4 hours after drug administration. No other medication or ventilator changes will be made during this time period outside of emergent changes in the setting of patient deterioration. We will continue to analyze the data in the event of emergent ventilator changes.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients at SBCH with confirmed COVID19 pneumonia (PCR + clinical signs/symptoms of lower respiratory disease)
* Patients currently on a ventilator
* Patients who meet the Berlin definition of ARDS
* Patients who have access to measure a mixed venous oxygen saturation (i.e., patients with an internal jugular central venous catheter)
* Patient and/or Legally Authorized Representative is willing/able to provide informed consent

Exclusion Criteria:

* As tadalafil is currently a FDA Class B1 medication, indicating that little information is available, pregnant women along with women who are actively breastfeeding will be excluded from this series.
* All patients under 18
* Patients who are routinely taking nitrate medications
* All patients using Tadalafil daily for pulmonary arterial hypertension (Note: patients using Tadalafil intermittently for erectile dysfunction may still participate in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Improvement in P:F ratio | Pre-medication, 30 minutes post medication, 4 hours post-medication
  Change in a patient's P:F ratio after medication administration
Improvement in oxygen saturation | Pre-medication, 30 minutes post medication, 4 hours post-medication
  Change in oxyhemoglobin as noted on an arterial blood gas sample after medication administration
Improvement in partial pressure of oxygen in the bloodstream | Pre-medication, 30 minutes post medication, 4 hours post-medication
  Change in oxygen partial pressure (aka PaO2) as noted on an arterial blood gas sample after medication administration

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers D, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Confirmation of the high cumulative incidence of thrombotic complications in critically ill ICU patients with COVID-19: An updated analysis. Thromb Res. 2020 Jul;191:148-150. doi: 10.1016/j.thromres.2020.04.041. Epub 2020 Apr 30. PMID 32381264
- [Background] Magro C, Mulvey JJ, Berlin D, Nuovo G, Salvatore S, Harp J, Baxter-Stoltzfus A, Laurence J. Complement associated microvascular injury and thrombosis in the pathogenesis of severe COVID-19 infection: A report of five cases. Transl Res. 2020 Jun;220:1-13. doi: 10.1016/j.trsl.2020.04.007. Epub 2020 Apr 15. PMID 32299776
- [Background] Keyaerts E, Vijgen L, Chen L, Maes P, Hedenstierna G, Van Ranst M. Inhibition of SARS-coronavirus infection in vitro by S-nitroso-N-acetylpenicillamine, a nitric oxide donor compound. Int J Infect Dis. 2004 Jul;8(4):223-6. doi: 10.1016/j.ijid.2004.04.012. PMID 15234326
- [Background] Akerstrom S, Mousavi-Jazi M, Klingstrom J, Leijon M, Lundkvist A, Mirazimi A. Nitric oxide inhibits the replication cycle of severe acute respiratory syndrome coronavirus. J Virol. 2005 Feb;79(3):1966-9. doi: 10.1128/JVI.79.3.1966-1969.2005. PMID 15650225
- [Background] Galie N, Brundage BH, Ghofrani HA, Oudiz RJ, Simonneau G, Safdar Z, Shapiro S, White RJ, Chan M, Beardsworth A, Frumkin L, Barst RJ; Pulmonary Arterial Hypertension and Response to Tadalafil (PHIRST) Study Group. Tadalafil therapy for pulmonary arterial hypertension. Circulation. 2009 Jun 9;119(22):2894-903. doi: 10.1161/CIRCULATIONAHA.108.839274. Epub 2009 May 26. PMID 19470885
- See also: Nu-Med Plus Closely Monitoring Outcomes on Two New Human Clinical Trials Using Inhaled Nitric Oxide in Treatment of COVID-19 — https://www.globenewswire.com/news-release/2020/03/25/2006042/0/en/Nu-Med-Plus-Closely-Monitoring-Outcomes-on-Two-New-Human-Clinical-Trials-Using-Inhaled-Nitric-Oxide-in-Treatment-of-COVID-19.html
- See also: A Pilot Study of Sildenafil in COVID-19 — https://clinicaltrials.gov/ct2/show/NCT04304313